CLINICAL TRIAL: NCT06650501
Title: Dabigatran vs. Apixaban, Edoxaban, or Rivaroxaban as Anti-thrombotic Therapy in Patients With S. Aureus Bacteremia: the DABI-SNAP Nested Randomized Controlled Trial
Brief Title: Dabigatran vs. Apixaban, Edoxaban, or Rivaroxaban as Anti-thrombotic Therapy in Patients With S. Aureus Bacteremia
Acronym: DABI-SNAP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emily McDonald (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Sponsor-Investigator, Emily McDonald, Associate Professor of Medicine and Staff Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-10900; 500464 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Staphylococcus Aureus Endocarditis; Staphylococcus Aureus Septicemia; Staphylococcus Aureus Bacteremia; Staphylococcus Aureus Bloodstream Infection; S. Aureus Bacteremia; S. Aureus Bloodstream Infection
Keywords: S. aureus bacteremia; S. aureus bloodstream infection; S. aureus endocarditis; Dabigatran; Edoxaban; Rivaroxaban; Apixaban
MeSH Terms: interventions — Dabigatran; apixaban; edoxaban; Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Change to Dabigatran (Experimental): Patients will have their anticoagulation changed to dabigatran at the monograph approved dose for the indication, bleeding risk, and renal function.
  Interventions: Drug: Dabigatran
- Continue current anticoagulant (Active Comparator): Patients will continue their currently prescribed apixaban, edoxaban, or rivaroxaban
  Interventions: Drug: Apixaban; Drug: edoxaban; Drug: Rivaroxaban

INTERVENTIONS:
Drug: Dabigatran — Patients will be assigned to change to dabigatran at the monograph approved dose for their indication, bleeding risk, and renal function.
  Arms: Change to Dabigatran
Drug: Apixaban — Patients will continue taking their currently prescribed apixaban, edoxaban, or rivaroxaban
  Arms: Continue current anticoagulant
Drug: edoxaban — Patients will continue taking their currently prescribed apixaban, edoxaban, or rivaroxaban
  Arms: Continue current anticoagulant
Drug: Rivaroxaban — Patients will continue taking their currently prescribed apixaban, edoxaban, or rivaroxaban
  Arms: Continue current anticoagulant

SUMMARY:
This is an open-label randomized controlled trial which will enroll patients with S. aureus bacteremia who are already taking oral anticoagulant medications (apixaban, edoxaban, or rivaroxaban) for an approved indication (stroke prevention in atrial fibrillation, prevention or treatment of venous thromboembolism). We will randomize patients to continue their existing medication or change to another medication (dabigatran) which is approved for the original indication.

Dabigatran is approved in many countries for the treatment or prevention of venous thromboembolism or preventing stroke in atrial fibrillation. Unlike the other medications listed above, dabigatran seems to have activity against S. aureus in the test tube, in animal models, and in a smaller randomized controlled trial. We wish to determine if changing to dabigatran will improve outcomes in S. aureus bacteremia in people who otherwise would have a reason to be taking it.

This study is an approved sub-study of The Staphylococcus aureus Network Adaptive Platform (SNAP) trial (NCT05137119).

If positive, this study will support a second RCT in people who do not currently have an indication for anticoagulation.

ELIGIBILITY:
The participant must meet all inclusion and exclusion criteria for the SNAP Platform (NCT05137119) and also the following inclusion and exclusion criteria:

Inclusion Criteria:

* Patient is taking (or will imminently start taking) an oral Xa inhibitor (e.g., apixaban, edoxaban, rivaroxaban) for: stroke prevention in atrial fibrillation, treatment or secondary prevention of deep venous thrombosis or pulmonary embolism, prevention of VTE in patients who have undergone elective total hip or total knee replacement surgery provided there are 30 or more days of planned treatment remaining at the time of enrolment.

Exclusion Criteria:

* Active bleeding as determine by the site investigator after discussion with the treating team (patient may remain eligible for up to 120 hours from platform entry if condition is resolved and antithrombotic therapy is resumed)
* Anticipated major cardiac surgery, neurosurgery, or spine surgery within the next 3 days
* Known pregnancy (with testing available for women with childbearing potential)
* Known use of dabigatran within last month
* Allergy to dabigatran
* Concomitant use of amiodarone, ketoconazole, rifampin, verapamil, clopidogrel, prasugrel, or ticagrelor
* eGFR < 30mL/minute calculated by Cockcroft-Gault equation using adjusted weight [patient may remain eligible for up to 120 hours from platform entry if acute kidney injury is resolved such that antithrombotic therapy can be safely resumed/prescribed]
* Off label use (e.g., metallic mechanical heart valve, left ventricular thrombus, antiphospholipid antibody syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Desirability of Outcome Ranking (DOOR) - an ordinal outcome with 5 levels defined:
  Rank 1 - Alive without complication Rank 2 - Alive with 1 complication Rank 3 - Alive with 2 complications Rank 4 - Alive with 3 complications Rank 5 - Dead
  Complications include:
  1. Clinical failure: Absence of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated.
  2. Infectious Complications: Including new endocarditis; new evidence of other deep metastatic foci (e.g., osteomyelitis or deep abscess); relapse of MRSA bacteremia after a patient has sterilized their initial blood cultures; readmission for subsequent care of S. aureus bacteremia; need for unplanned source control procedures
  3. Serious adverse drug event (Common Terminology Criteria class 4) due to study drug OR adverse drug event (classes 1-3) leading to discontinuation of the study drug

SECONDARY OUTCOMES:
Clinical failure | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as the absence of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated for its treatment.
Serious Adverse Event or Adverse Event Leading to Discontinuation | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as a serious adverse drug event (Common Terminology Criteria for Adverse Events (CTCAE) class 4) presumed due to study drug OR adverse drug event (CTCAE classes 1-3) leading to discontinuation of the study drug
All cause mortality | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Death from any cause
Infectious Complications | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as change in therapy for inadequate clinical response; new endocarditis; new evidence of other deep metastatic foci (e.g., osteomyelitis or deep abscess); relapse of MRSA bacteremia after a patient has sterilized their initial blood cultures; readmission for subsequent care of S. aureus bacteremia; need for unplanned source control procedures. New implies that the complication was not suspected at enrollment and is not a function of delay to diagnostic testing.
Clinically relevant major bleeding | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  This will be defined according to the criteria of the International Society on Thrombosis and Haemostasis as one or more of the following: fatal bleeding; symptomatic bleeding in a critical area or organ (including hemorrhagic stroke); bleeding that causes a fall in hemoglobin level of ≥20 g/L; or bleeding that requires a transfusion of 2 or more units of whole blood or red cells. For bleeds into non-critical areas, we will also record the site of bleeding.
Clinically relevant venous thromboembolic events | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  This will be defined as an acute objectively confirmed deep vein thrombosis (upper extremity, lower extremity, other such as portal vein, cerebral vein, splanchnic vein) and/or segment or proximal pulmonary embolism, which is symptomatic and/or necessitates specific treatment. Below knee DVT and superficial thrombophlebitis are not included. Pulmonary embolism needs to be, segmental or proximal. Subsegmental pulmonary embolisms are not included as they have poor interrater reliability and may represent artefact in up to 50% of cases.
Clinically relevant stroke | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Stroke is defined as the acute onset of focal neurological dysfunction caused by brain, spinal cord, or retinal vascular injury because of infarction (ischemia). Ideally, at least one of the following should be present to confirm the diagnosis of stroke: confirmation by neurology, stroke specialist, or neurosurgical specialist, brain imaging (e.g., CT scan, MRI scan, or cerebral vessel angiography compatible with acute ischemia). If the acute focal signs represent a worsening of a previous deficit, these signs must persist for more than 24 hours and be accompanied by an appropriate new MRI or CT scan finding. In the absence of neuroimaging, a staff neurologist consult which makes the diagnosis of stroke will be considered.
Clinically relevant acute myocardial infarction | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Patients with S. aureus bacteremia often have substantial physiological stresses which can be associated with rises in cardiac troponin (demand ischemia). For the purposes of this outcome, acute myocardial infarction is captured as a type 1 myocardial infarction: detection of rise and/or fall of cardiac biomarkers with at least one value above the 99th percentile of the upper reference limit together with evidence of myocardial ischemia. For the purposes of this pragmatic trial, such a myocardial infarction will be inferred from the opinions of the staff cardiologist, intensivist, or general internal medicine specialist. The peak troponin value will be recorded, and a redacted copy of the relevant consultant's note and ECGs will be uploaded for audit.
Clinically relevant arterial thromboembolic event | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Clinical history compatible with sudden worsening of end organ or limb perfusion and confirmation by imaging (e.g., CT angiography, arterial doppler) or need for urgent surgery or thrombolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Emily G McDonald, MD MSC, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre (Royal Victoria Hospital and Montreal General Hospital), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
This statement supersedes any such statement in NCT05137119.
  For DABI-SNAP, we will provide deidentified individual patient data required to replicate the main manuscript's tables and analyses.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting 1 year after the publication of the main trial manuscript for up to 7 years.
Access Criteria: Researchers will need to request the data from the corresponding author of the main trial manuscript with an accompanying written proposal for the secondary analysis. Once approved by the trial steering committee, a data sharing agreement will be signed by the responsible parties and the deidentified data set will be provided via a secure transmission.

REFERENCES:
- [Background] Lerche CJ, Christophersen LJ, Goetze JP, Nielsen PR, Thomsen K, Enevold C, Hoiby N, Jensen PO, Bundgaard H, Moser C. Adjunctive dabigatran therapy improves outcome of experimental left-sided Staphylococcus aureus endocarditis. PLoS One. 2019 Apr 19;14(4):e0215333. doi: 10.1371/journal.pone.0215333. eCollection 2019. PMID 31002679
- [Background] Butt JH, Fosbol EL, Verhamme P, Gerds TA, Iversen K, Bundgaard H, Bruun NE, Larsen AR, Petersen A, Andersen PS, Skov RL, Gislason GH, Torp-Pedersen C, Kober L, Olesen JB. Dabigatran and the Risk of Staphylococcus aureus Bacteremia: A Nationwide Cohort Study. Clin Infect Dis. 2021 Aug 2;73(3):480-486. doi: 10.1093/cid/ciaa661. PMID 32478836
- [Background] Vanassche T, Verhaegen J, Peetermans WE, VAN Ryn J, Cheng A, Schneewind O, Hoylaerts MF, Verhamme P. Inhibition of staphylothrombin by dabigatran reduces Staphylococcus aureus virulence. J Thromb Haemost. 2011 Dec;9(12):2436-46. doi: 10.1111/j.1538-7836.2011.04529.x. PMID 22040101
- [Background] Vanassche T, Verhaegen J, Peetermans WE, Hoylaerts MF, Verhamme P. Dabigatran inhibits Staphylococcus aureus coagulase activity. J Clin Microbiol. 2010 Nov;48(11):4248-50. doi: 10.1128/JCM.00896-10. Epub 2010 Sep 1. PMID 20810780
- [Background] Peetermans M, Liesenborghs L, Peerlinck K, Wijngaerden EV, Gheysens O, Goffin KE, Hoylaerts MF, Jacquemin M, Verhaegen J, Peetermans WE, Verhamme P, Vanassche T; Staphylothrombin Investigators. Targeting Coagulase Activity in Staphylococcus aureus Bacteraemia: A Randomized Controlled Single-Centre Trial of Staphylothrombin Inhibition. Thromb Haemost. 2018 May;118(5):818-829. doi: 10.1055/s-0038-1639586. Epub 2018 Apr 3. PMID 29614521
- [Background] Tong SYC, Mora J, Bowen AC, Cheng MP, Daneman N, Goodman AL, Heriot GS, Lee TC, Lewis RJ, Lye DC, Mahar RK, Marsh J, McGlothlin A, McQuilten Z, Morpeth SC, Paterson DL, Price DJ, Roberts JA, Robinson JO, van Hal SJ, Walls G, Webb SA, Whiteway L, Yahav D, Davis JS; Staphylococcus aureus Network Adaptive Platform (SNAP) Study Group. The Staphylococcus aureus Network Adaptive Platform Trial Protocol: New Tools for an Old Foe. Clin Infect Dis. 2022 Nov 30;75(11):2027-2034. doi: 10.1093/cid/ciac476. PMID 35717634
- [Derived] McDonald EG, Cheng MP, Davis JS, Goodman AL, Lawler PR, Marsh J, Mertz D, Paul M, Rodriguez-Bano J, Siegal DM, Tong SY, Walls G, Lee TC; SNAP Global Trial Steering Committee. Is there a role for anticoagulation with dabigatran in S. aureus bacteremia? Protocol for the adjunctive treatment domain of the Staphylococcus aureus Network Adaptive Platform (SNAP) randomised controlled trial. BMJ Open. 2025 Dec 12;15(12):e107493. doi: 10.1136/bmjopen-2025-107493. PMID 41387009
- See also: Website for the S. aureus Network Adaptive Platform Trial (SNAP) — https://www.snaptrial.com.au/